CLINICAL TRIAL: NCT03474809
Title: A Multicenter, Device Clinical Study for the Early Diagnostic of Sepsis and Potential Impact on Antibiotic Management Based on Serial Pancreatic Stone Protein (PSP) Measured Using the AbioScope in Critically Ill Patients at High Risk of Sepsis.
Brief Title: Early Diagnostic of Sepsis and Potential Impact on Antibiotic Management Based on Serial.Pancreatic Stone Protein (PSP) Measured Using the AbioScope.
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-PSP-001
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sepsis
Keywords: Sepsis, PSP, Abionic
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood sampling — Daily blood samples which will be taken for the PSP measurement using the AbioScope as well as another daily sample taken for central analysis of biomarkers of inflammation, infection and/or sepsis (including but not limited to C-reactive protein [CRP] and Procalcitonin [PCT]).

SUMMARY:
The main purpose of this study is to compare the early detection of sepsis and the decision, by the Investigator to start or not, or to change, antibiotics in Intensive Care Unit (ICU) patients at high risk of sepsis, based on standard of care (clinical, laboratory and imaging data but not on PSP values), as well as timing of antibiotic de-escalation versus the the retrospective assessment (i.e., at the end of the study) of a First Endpoint Adjudication Committee (EAC) which is aware of the clinical data and of the PSP values but not of the Investigator's decision(s), and of the retrospective assessment of a Second Endpoint Adjudication Committee which is only aware of the PSP values.

This study will follow the site's routine clinical practice for the diagnostic, assessment and treatment of the enrolled patients, with the exception of daily blood samples which will be taken for the PSP measurement using the AbioScope as well as another daily sample taken for central analysis of biomarkers of inflammation, infection and/or sepsis (including but not limited to C-reactive protein [CRP] and Procalcitonin [PCT]).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years)
2. Requiring ICU management
3. At high risk of sepsis (septic patients are excluded)
4. Expected ICU stay for more than 4 days
5. Have provided written informed consent or consent is given by the patient's legally designated representative.

Exclusion Criteria:

1. Patient expected to die within 48 hours of admission to ICU
2. Patient suffering from or known acute or chronic pancreatitis, pancreatic cancer or admitted after pancreatectomy, but if a patient develops any pancreatic disease during the IUC stay he/she will remain in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients at high risk of sepsis admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the performance of serial PSP values measured using the AbioScope. | Day 1 to Day 30, or until discharge from ICU
  i) To assess the performance of serial PSP values measured using the AbioScope in the early detection of sepsis in ICU patients at high risk of developing sepsis.

CONTACTS AND LOCATIONS:
Locations (14):
- France (4):
  - CH Le Mans, Service de Réanimation Médico Chirurgicale & USC, Le Mans
  - CHU Limoges, Réanimation Polyvalente, Limoges
  - CH Lyon-Sud, Services de soins critiques, Pierre-Bénite
  - Hôpital Bretonneau, CHU de Tours, Médecine Intensive - Réanimation, Tours
- Italy (4):
  - Ospedale Santa Maria della Misericordia, Terapia Intensiva, Perugia
  - Ospedale Santa Maria delle Croci, Terapia Intensiva, Ravenna
  - Ospedale Infermi, Dept Anesthesia and ICU, Rimini
  - Ospedale San Giovanni Bosco, Servizio Anestesia e Rianimazione, Torino
- Switzerland (3):
  - Bern University Hospital, Universitätsklinik für Intensivmedizin, Bern
  - Hopitaux Universitaires de Genève, Service des soins intensifs, Département APSI, Geneva
  - Centre Hospitalier Universitaire Vaudois, Service of Adult Intensive Care, Lausanne
- United Kingdom (3):
  - Royal Surrey County Hospital, Intensive Care Medicine, Guildford
  - University College London Hospitals, Anaesthetics Department, London
  - Guy's & St Thomas' Hospital, Department of Critical Care, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pugin J, Daix T, Pagani JL, Morri D, Giacomucci A, Dequin PF, Guitton C, Que YA, Zani G, Brealey D, Lepape A, Creagh-Brown B, Wyncoll D, Silengo D, Irincheeva I, Girard L, Rebeaud F, Maerki I, Eggimann P, Francois B. Serial measurement of pancreatic stone protein for the early detection of sepsis in intensive care unit patients: a prospective multicentric study. Crit Care. 2021 Apr 20;25(1):151. doi: 10.1186/s13054-021-03576-8. PMID 33879189